CLINICAL TRIAL: NCT01934946
Title: Effectiveness of Post Acute Rehabilitation Care for Hip Fracture
Brief Title: Rehabilitation Care for Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, MUJUNG KAO, Director, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCHIRB-1020430
Record Dates: First submitted 2013-08-22; First posted 2013-09-04 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Hip Fracture
Keywords: hip fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- comprehensive rehabilitation 10 days (Experimental): comprehensive rehabilitation PT OT once per day for 10 times within 14 days hospitalization
  Interventions: Other: comprehensive rehabilitation
- home rehabilitation (Placebo Comparator): home rehabilitation 6 times of PT home visit within 3 months after discharge
  Interventions: Other: home rehabilitation

INTERVENTIONS:
Other: comprehensive rehabilitation — received 14 days hospitalization for comprehensive rehabilitation
  Arms: comprehensive rehabilitation 10 days
Other: home rehabilitation — 6 times home rehabilitation services within 3 months
  Arms: home rehabilitation

SUMMARY:
Purpose: Hip fracture is a common disease on elderly. They become disabled easily if no adequate rehabilitation was given. The aim of the study is to compare the effectiveness of different types of post acute rehabilitation care for hip fracture.

DETAILED DESCRIPTION:
Method: This study will recruit 150 peoples with hip fracture from hospitals in Taipei from Jan 1, 2014 to Dec 31, 2014. The subjects from wards are randomly divided into group A, B and Group C. Each group includes 50 cases of hip fracture. Group C received 14 days hospitalization for comprehensive rehabilitation and 6 times home rehabilitation services within 3 months; Group B received 14 days hospitalization for comprehensive rehabilitation and Group A was control group.

ELIGIBILITY:
Inclusion Criteria:

1. more than 60 years old,
2. hip fracture s/p within 3 months,
3. potential for rehabilitation.

Exclusion Criteria:

1. Active infection, such as pneumonia, UTI, osteomyelitis, wound infection
2. Other uncontrolled medical condition, such as, dyspnea on exertion, acute renal failure, acute coronary syndrome, acute heart failure, uncontrolled diabetes, active malignancy, DVT, possibility of pulmonary embolism, acute psychosis
3. No caregiver
4. No potential for rehabilitation, such as severe dementia, poor cognition, poor cooperation and motivation, poor family support
5. ESRD on Hemodialysis

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 2 weeks and 3 months after intervention
  change

SECONDARY OUTCOMES:
Barthel Activity of Daily Living | 2 weeks , 3 months after intervention
  change

OTHER OUTCOMES:
Harris Hip Score | 2 weeks , 3 months after intervention
  change

CONTACTS AND LOCATIONS:
Overall Officials: MUJUNG KAO, MD, Principal Investigator — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan